CLINICAL TRIAL: NCT01563029
Title: A Dose-ranging Study of Fluticasone Furoate (FF) Inhalation Powder in Children Aged 5-11 Years With Asthma
Brief Title: A Dose-ranging Study of Fluticasone Furoate (FF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 106855
Record Dates: First submitted 2012-03-15; First posted 2012-03-26 (Estimated); Results first posted 2015-04-27 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Active Comparator): Fluticasone Furoate 100mcg inhalation powder once daily in the evening ICS powder
  Interventions: Drug: Fluticasone Furoate
- Arm 2 (Active Comparator): Fluticasone Furoate 50mcg inhalation powder once daily in the evening ICS powder
  Interventions: Drug: Fluticasone Furoate
- Arm 3 (Active Comparator): Fluticasone Furoate 25mcg inhalation powder once daily in the evening ics powder
  Interventions: Drug: Fluticasone Furoate
- Arm 4 (Active Comparator): Fluticasone Propionate 100mcg inhalation powder twice daily ICS powder
  Interventions: Drug: Fluticasone Propionate
- Arm 5 (Placebo Comparator): Placebo inhalation powder once daily in the evening Placebo powder
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone Furoate — current asthma medicine
  Arms: Arm 1; Arm 2; Arm 3
Drug: Fluticasone Propionate — Fluticasone propionate
  Arms: Arm 4
Drug: Placebo — placebo
  Arms: Arm 5

SUMMARY:
This is a Phase IIb, multi-centre, stratified, randomised, double-blind, double-dummy, parallel-group, placebo and active controlled study in children aged 5-11 years with persistent uncontrolled asthma. Subjects meeting all of the inclusion criteria and none of the exclusion criteria at the screening visit (Visit 1) will enter a four week run-in period during which time they will continue their current medications. Visit 2 will occur two weeks into the run-in period to allow a review of compliance with daily diary and run-in medication. At Visit 3 (end of run-in/randomization visit), subjects meeting the eligibility criteria who remain uncontrolled despite baseline therapy will be stratified based on pre screening inhaled corticosteroid (ICS) use. Once stratified, subjects will be randomised to the treatment phase of the study where they will receive one of five treatments for 12 weeks. Approx 1200 subjects ages 5 to 11 will be screened to achieve 575 randomized for a total of 115 randomized/evaluable subjects per treatment arm. Subjects will attend on-treatment visits at 2, 4, 8 and 12 weeks (Visits 4, 5, 6 and 7 respectively). A follow-up contact will be performed one week after completing study medication. All subjects must attempt spirometry measurements at Visits 1 and 3. For all subjects, a timed 24-hour urine collection for urinary cortisol and creatinine excretion will be performed prior to randomization at Visit 2 and within 7 days prior to Visit 7. All subjects must perform PEF daily between visits 1 and 7. The primary endpoint will be change from baseline in pre-dose (i.e. dosing trough) PM PEF from patient hand held electronic daily diary at Endpoint (Endpoint is defined as the mean over the last 7 days of treatment). Safety assessments include adverse events, oropharyngeal examinations, clinical chemistry, urinary cortisol, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from at least one parent/ legal guardian to take part in the study.:
* Diagnosis of asthma
* pre-bronchodilator PEF between ≥50% to ≤90% of their best post-bronchodilator value
* Receiving therapy of short acting beta-agonist (SABA) alone, LTM, or ICS (total daily dose <FP 200mcg or equivalent)Exclusion :

Exclusion Criteria:

* history of life-threatening asthma
* history of asthma exacerbation for asthma within 6 months prior to screening.
* Culture-documented or suspected bacterial or viral infection
* significant abnormality or medical condition
* Present use of any tobacco products

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 597 (Actual)
Dates: Start 2012-03-28 (Actual); Primary Completion 2014-09-24 (Actual); Study Completion 2014-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (118):
- United States (36):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Costa Mesa, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Eagle, Idaho
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Shiloh, Illinois
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, Corning, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, South Burlington, Vermont
- Bulgaria (3):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
- GSK Investigational Site, Tbilisi, Georgia
- Germany (17):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Berchtesgaden, Bavaria
  - GSK Investigational Site, Rosenheim, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Niedernhausen, Hesse
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Hamm, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Telgte, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Neuhaus am Rennweg, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Japan (10):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Wakayama
- Latvia (3):
  - GSK Investigational Site, Daugavpils
  - GSK Investigational Site, Rēzekne
  - GSK Investigational Site, Riga
- Mexico (6):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Morelia, Michoacán
  - GSK Investigational Site, Villahermosa, Tabasco
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- Peru (4):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, San Borja, Lima region
  - GSK Investigational Site, San Miguel, Lima region
  - GSK Investigational Site, Lima
- Philippines (2):
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
- Poland (8):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Tarnów
- GSK Investigational Site, Hato Rey, Puerto Rico, Puerto Rico
- Russia (8):
  - GSK Investigational Site, Blagoveshchensk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Murmansk
  - GSK Investigational Site, Novokuznetsk
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
- South Africa (3):
  - GSK Investigational Site, Panorama, Western Province
  - GSK Investigational Site, CapeTown
  - GSK Investigational Site, Middelburg
- Sweden (6):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Kungsbacka
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
  - GSK Investigational Site, Visby
- Ukraine (10):
  - GSK Investigational Site, Chernivtsi
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kherson
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Luhansk
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Yevpatoriia
  - GSK Investigational Site, Zaporizhia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Oliver AJ, Covar RA, Goldfrad CH, Klein RM, Pedersen SE, Sorkness CA, Tomkins SA, Villaran C, Grigg J. Randomized Trial of Once-Daily Fluticasone Furoate in Children with Inadequately Controlled Asthma. J Pediatr. 2016 Nov;178:246-253.e2. doi: 10.1016/j.jpeds.2016.08.010. Epub 2016 Sep 9. PMID 27622699
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 106855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1540 participants were screened, 596 participants were randomized, and 593 participants comprise the Intent to Treat Population which include all participants who received at least one dose of study treatment. Participants were stratified at randomization according to their prior inhaled corticosteroid (ICS) use.
Pre-assignment Details: Participants who met the eligibility criteria at screening (Visit 1) entered a 4-week Run-in Period during which they continued their existing medications. Participants who met the randomization criteria (remained uncontrolled despite baseline therapy) at Visit 3 were randomized to 1 of 5 treatment arms for 12 weeks followed by a 1-week follow-up.
Groups:
- Placebo: Participants received placebo once daily (OD) in the evening via a dry powder inhaler (DPI) and placebo twice daily (BID), once in the morning and once in the evening via a separate DPI for 12 weeks. Participants were also provided albuterol/salbutamol inhalation aerosol via metered dose inhaler (MDI) to be used as rescue medication as determined by the investigator.
- FF 25 µg OD: Participants received fluticasone furoate (FF) 25 micrograms (µg) OD in the evening via a DPI and placebo BID, once in the morning and once in the evening via a separate DPI for 12 weeks. Participants were also provided albuterol/salbutamol inhalation aerosol via metered dose inhaler (MDI) to be used as rescue medication as determined by the investigator.
- FF 50 µg OD: Participants received FF 50 µg OD in the evening via a DPI and placebo BID, once in the morning and once in the evening via a separate DPI for 12 weeks. Participants were also provided albuterol/salbutamol inhalation aerosol via metered dose inhaler (MDI) to be used as rescue medication as determined by the investigator.
- FF 100 µg OD: Participants received FF 100 µg OD in the evening via a DPI and placebo BID, once in the morning and once in the evening via a separate DPI for 12 weeks. Participants were also provided albuterol/salbutamol inhalation aerosol via metered dose inhaler (MDI) to be used as rescue medication as determined by the investigator.
- FP 100 µg BID: Participants received fluticasone propionate (FP) 100 µg BID, once in the morning and once in the evening via a DPI and placebo OD in the evening via a separate DPI for 12 weeks. Participants were also provided albuterol/salbutamol inhalation aerosol via metered dose inhaler (MDI) to be used as rescue medication as determined by the investigator.
Period: Overall Study
Arm/Group | Placebo | FF 25 µg OD | FF 50 µg OD | FF 100 µg OD | FP 100 µg BID
Started | 119 | 118 | 120 | 118 | 118
Completed | 66 | 94 | 87 | 85 | 89
Not Completed | 53 | 24 | 33 | 33 | 29
Not completed — Adverse Event | 1 | 0 | 1 | 2 | 1
Not completed — Lack of Efficacy | 42 | 16 | 23 | 21 | 19
Not completed — Protocol Violation | 1 | 2 | 3 | 1 | 3
Not completed — Protocol defined stopping criteria | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1 | 1
Not completed — Physician Decision | 3 | 5 | 2 | 4 | 2
Not completed — Withdrawal by Subject | 4 | 1 | 3 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FF 25 µg OD | FF 50 µg OD | FF 100 µg OD | FP 100 µg BID | Total
Number analyzed (Participants) | 119 | 118 | 120 | 118 | 118 | 593
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.0 (1.91) | 7.9 (2.08) | 8.4 (1.62) | 7.8 (2.04) | 7.9 (1.87) | 8.0 (1.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 41 | 46 | 48 | 39 | 223
  Male | 70 | 77 | 74 | 70 | 79 | 370
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 4 | 4 | 7 | 8 | 7 | 30
  American Indian or Alaskan Native | 24 | 17 | 16 | 17 | 21 | 95
  Asian -Central/South Asian Heritage | 1 | 0 | 1 | 0 | 0 | 2
  Asian - Japanese Heritage | 7 | 7 | 5 | 2 | 7 | 28
  White - Arabic/North African Heritage | 1 | 2 | 0 | 1 | 0 | 4
  White - White/Caucasian/European Heritage | 47 | 55 | 51 | 51 | 43 | 247
  Mixed Race | 35 | 33 | 40 | 39 | 40 | 187

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Pre-dose Morning (AM) Peak Expiratory Flow (PEF) From Participant Electronic Daily Diary Averaged Over the 12-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. The best of three measurements was recorded. Change from Baseline was calculated as the value of the averaged daily AM PEF over the 12-week Treatment Period minus the Baseline value. The Baseline PEF value is defined as the average of the last 7 days of the Run-in Period. Statistical analysis was performed using an analysis of covariance (ANCOVA) model with covariates of Baseline AM PEF, actual pre-screening inhaled corticosteroid (ICS) use, region, sex, age, and treatment. Particpants analyzed included those who have PEF data for at least 2 non-missing days in the Baseline week prior to randomisation and at least 2 non-missing days after randomisation.
Time Frame: Baseline; Week 1 up to Week 12
Population: ITT Population: participants randomized to treatment who received at least 1 dose of study medication. Only participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Deviation); unit: Liters per minute (L/min)
Groups:
- Average of FF 50 µg OD and FF 100 µg OD: All participants who received FF 100 µg OD in the evening via a DPI and placebo BID, once in the morning and once in the evening via a separate DPI for 12 weeks and all participants who FF 50 µg OD in the evening via a DPI and placebo BID, once in the morning and once in the evening via a separate DPI for 12 weeks. Participants were also provided albuterol/salbutamol inhalation aerosol via metered dose inhaler (MDI) to be used as rescue medication as determined by the investigator.
Arm/Group | Placebo | FF 25 µg OD | FF 50 µg OD | FF 100 µg OD | FP 100 µg BID | Average of FF 50 µg OD and FF 100 µg OD
Number analyzed (Participants) | 119 | 117 | 118 | 118 | 117 | 236
Liters per minute (L/min) | 3.3 (2.63) | 21.9 (2.66) | 22.8 (2.65) | 15.8 (2.64) | 17.3 (2.64) | 19.3 (1.86)
Statistical Analysis 1: Comparison: Placebo vs Average of FF 50 µg OD and FF 100 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Gate-keeper analysis; Mean Difference (Final Values) = 16.0, 95% CI 2-sided [9.6 to 22.4]
Statistical Analysis 2: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 12.5, 95% CI 2-sided [5.1 to 19.8] — Inference for FF 100 μg versus (vs) placebo and FF 50 ug versus placebo was dependent upon statistical significance (SS) having first been achieved for the average of the higher two doses of FF (FF 100 ug and 50 ug ) versus placebo comparison
Statistical Analysis 3: Comparison: Placebo vs FF 50 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 19.5, 95% CI 2-sided [12.1 to 26.9] — Inference for FF 100 µg versus (vs) placebo and FF 50 ug versus placebo was dependent upon statistical significance (SS) having first been achieved for the average of the higher two doses of FF (FF 100 ug and 50 ug ) versus placebo comparsion
Statistical Analysis 4: Comparison: Placebo vs FF 25 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 18.6, 95% CI 2-sided [11.3 to 26.0] — Inference for FF 25 ug versus placebo was dependent upon statistical significance (SS) having first been achieved for both the FF 100 ug versus placebo comparison and the FF 50 ug versus placebocomparison
Statistical Analysis 5: Comparison: Placebo vs FP 100 µg BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = 14.0, 95% CI 2-sided [6.7 to 21.4]

2. Secondary Outcome: Change From Baseline in Evening Clinic Visit Trough (Pre-bronchodilator and Pre-dose) Forced Expiratory Volume in One Second (FEV1) at the End of the 12-week Treatment Period in Children Who Could Perform the Maneuver
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 is defined as a pre-dose FEV1 measurement taken at a clinic visit while still on treatment. Change from Baseline was calculated as the Week 12 trough FEV1 value minus the Baseline value. The Baseline FEV1 value is defined as the value at Visit 3 (randomization). The analysis was performed using an ANCOVA model with covariates of Baseline trough FEV1, region, actual pre-screening ICS use, sex, age, and treatment. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement at scheduled clinic visits was used to impute the missing measurements. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline, Week 12
Population: ITT Population. Only participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF 25 µg OD | FF 50 µg OD | FF 100 µg OD | FP 100 µg BID
Number analyzed (Participants) | 102 | 96 | 112 | 96 | 102
Liters | 0.128 (0.0264) | 0.254 (0.0272) | 0.150 (0.0252) | 0.162 (0.0272) | 0.192 (0.0262)
Statistical Analysis 1: Comparison: Placebo vs FF 25 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.126, 95% CI 2-sided [0.051 to 0.201]
Statistical Analysis 2: Comparison: Placebo vs FF 50 µg OD; Test type: Superiority or Other; p = 0.551, ANCOVA; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.050 to 0.094]
Statistical Analysis 3: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p = 0.379, ANCOVA; Mean Difference (Final Values) = 0.033, 95% CI 2-sided [-0.041 to 0.108]
Statistical Analysis 4: Comparison: Placebo vs FP 100 µg BID; Test type: Superiority or Other; p = 0.089, ANCOVA; Mean Difference (Final Values) = 0.064, 95% CI 2-sided [-0.010 to 0.137]

3. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour Periods During the 12-week Treatment Period
Description: The number of inhalations of rescue albuterol/salbutamol aerosol (medication used to relieve symptoms immediately) used during the day and night) was recorded by the participants in a daily diary. A 24-hour (hr) period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered as rescue free. The Baseline rescue-free value was defined as the percentage of rescue-free 24-hr periods from the last 7 days of the Run-in Period. Change from Baseline was calculated as the average value during the 12-week Treatment Period minus the value at Baseline. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, actual pre-screening ICS use, age, and treatment.
Time Frame: Baseline; Week 1 up to Week 12
Population: ITT Population. Only participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | Placebo | FF 25 µg OD | FF 50 µg OD | FF 100 µg OD | FP 100 µg BID
Number analyzed (Participants) | 119 | 117 | 118 | 118 | 117
Percentage of rescue-free 24-hr periods | 16.5 (3.01) | 24.9 (3.03) | 26.3 (3.03) | 28.7 (3.02) | 22.7 (3.01)
Statistical Analysis 1: Comparison: Placebo vs FF 25 µg OD; Test type: Superiority or Other; p = 0.050, ANCOVA; Mean Difference (Final Values) = 8.4, 95% CI 2-sided [0.0 to 16.9]
Statistical Analysis 2: Comparison: Placebo vs FF 50 µg OD; Test type: Superiority or Other; p = 0.023, ANCOVA; Mean Difference (Final Values) = 9.8, 95% CI 2-sided [1.3 to 18.2]
Statistical Analysis 3: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = 12.2, 95% CI 2-sided [3.8 to 20.5]
Statistical Analysis 4: Comparison: Placebo vs FP 100 µg BID; Test type: Superiority or Other; p = 0.143, ANCOVA; Mean Difference (Final Values) = 6.2, 95% CI 2-sided [-2.1 to 14.6]

4. Secondary Outcome: Change From Baseline in Daily Evening (PM) PEF Averaged Over the 12-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline was calculated as the value of the averaged daily PM PEF over the 12-week Treatment Period (at Week 12) minus the Baseline value. The Baseline PEF value is defined as the average of the last 7 days of the Run-in Period. Statistical analysis was performed using ANCOVA model with covariates of Baseline, actual pre-screening ICS use, region, sex, age, and treatment. Particpants analyzed included those who have PEF data for at least 2 non-missing days in the Baseline week prior to randomisation and at least 2 non-missing days after randomisation.
Time Frame: Baseline; Week 1 up to Week 12
Population: ITT Population. Only participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: liters per minute (L/min)
Arm/Group | Placebo | FF 25 µg OD | FF 50 µg OD | FF 100 µg OD | FP 100 µg BID
Number analyzed (Participants) | 119 | 117 | 119 | 118 | 117
liters per minute (L/min) | 5.1 (2.76) | 16.3 (2.81) | 18.5 (2.77) | 13.5 (2.78) | 13.1 (2.77)
Statistical Analysis 1: Comparison: Placebo vs FF 25 µg OD; Test type: Superiority or Other; p = 0.005, ANCOVA; Mean Difference (Final Values) = 11.2, 95% CI 2-sided [3.4 to 19.0]
Statistical Analysis 2: Comparison: Placebo vs FF 50 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 13.4, 95% CI 2-sided [5.7 to 21.1]
Statistical Analysis 3: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p < 0.033, ANCOVA; Mean Difference (Final Values) = 8.4, 95% CI 2-sided [0.7 to 16.1]
Statistical Analysis 4: Comparison: Placebo vs FP 100 µg BID; Test type: Superiority or Other; p = 0.042, ANCOVA; Mean Difference (Final Values) = 8.0, 95% CI 2-sided [0.3 to 15.7]

5. Secondary Outcome: Change From Baseline in PM PEF Over the Last 7 Days of the Treatment Period (Week 12)
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline in PM PEF was calculated as the value over the last 7 days of the Treatment Period minus the Baseline value. The Baseline PEF value is defined as the average of the last 7 days of the Run-in Period. Statistical analysis was performed using ANCOVA model with covariates of Baseline, actual pre-screening ICS use, region, sex, age, and treatment. The LOCF method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurements.
Time Frame: Baseline; Week 12
Population: ITT Population. Only participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | FF 25 µg OD | FF 50 µg OD | FF 100 µg OD | FP 100 µg BID
Number analyzed (Participants) | 119 | 117 | 118 | 118 | 117
L/min | 5.0 (3.75) | 16.2 (3.80) | 18.2 (3.77) | 11.0 (3.76) | 11.3 (3.75)
Statistical Analysis 1: Comparison: Placebo vs FF 25 µg OD; Test type: Superiority or Other; p = 0.037, ANCOVA; Mean Difference (Final Values) = 11.2, 95% CI 2-sided [0.7 to 21.7]
Statistical Analysis 2: Comparison: Placebo vs FF 50 µg OD; Test type: Superiority or Other; p = 0.014, ANCOVA; Mean Difference (Final Values) = 13.1, 95% CI 2-sided [2.6 to 23.6]
Statistical Analysis 3: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p = 0.266, ANCOVA; Mean Difference (Final Values) = 5.9, 95% CI 2-sided [-4.5 to 16.3]
Statistical Analysis 4: Comparison: Placebo vs FP 100 µg BID; Test type: Superiority or Other; p = 0.242, ANCOVA; Mean Difference (Final Values) = 6.2, 95% CI 2-sided [-4.2 to 16.6]

6. Secondary Outcome: Change From Baseline in AM PEF Over the Last 7 Days of the Treatment Period (Week 12)
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline in AM PEF was calculated as the value over the last 7 days of the Treatment Period minus the Baseline value. The Baseline PEF value is defined as the average of the last 7 days of the Run-in Period. Statistical analysis was performed using ANCOVA model with covariates of Baseline, pre-screening ICS use, region, sex, age, and treatment. The LOCF method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurements.
Time Frame: Baseline; Week 12
Population: ITT Population. Only participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | FF 25 µg OD | FF 50 µg OD | FF 100 µg OD | FP 100 µg BID
Number analyzed (Participants) | 119 | 117 | 118 | 118 | 117
L/min | 2.7 (3.81) | 23.3 (3.85) | 20.6 (3.83) | 14.2 (3.82) | 19.3 (3.82)
Statistical Analysis 1: Comparison: Placebo vs FF 25 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 20.6, 95% CI 2-sided [10.0 to 31.3]
Statistical Analysis 2: Comparison: Placebo vs FF 50 µg OD; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = 17.9, 95% CI 2-sided [7.2 to 28.6]
Statistical Analysis 3: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p = 0.033, ANCOVA; Mean Difference (Final Values) = 11.5, 95% CI 2-sided [0.9 to 22.1]
Statistical Analysis 4: Comparison: Placebo vs FP 100 µg BID; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = 16.7, 95% CI 2-sided [6.0 to 27.3]

7. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour Periods During the 12-week Treatment Period
Description: Asthma symptoms were recorded in a daily eDairy by the participants every day in the morning and evening before taking any rescue or study medication and before the PEF measurement. A 24-hour (hr) period in which a participant's responses to both the morning and evening assessments indicated no symptoms was considered to be symptom free. The Baseline symptom-free value is defined as the percentage of symptom free 24-hr periods in the last 7 days of the run-in period. Change from Baseline was calculated as the averaged value during the 12-week Treatment Period minus the Baseline value. The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, actual pre-screening ICS use, age, and treatment group.
Time Frame: Baseline; Week 1 up to Week 12
Population: ITT Population. Only participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hr periods
Arm/Group | Placebo | FF 25 µg OD | FF 50 µg OD | FF 100 µg OD | FP 100 µg BID
Number analyzed (Participants) | 119 | 117 | 119 | 118 | 117
Percentage of symptom-free 24-hr periods | 19.0 (2.90) | 21.0 (2.92) | 24.7 (2.90) | 22.9 (2.91) | 22.0 (2.91)
Statistical Analysis 1: Comparison: Placebo vs FF 25 µg OD; Test type: Superiority or Other; p = 0.619, ANCOVA; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-6.1 to 10.2]
Statistical Analysis 2: Comparison: Placebo vs FF 50 µg OD; Test type: Superiority or Other; p = 0.161, ANCOVA; Mean Difference (Final Values) = 5.8, 95% CI [-2.3 to 13.9]
Statistical Analysis 3: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p = 0.340, ANCOVA; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [-4.1 to 12.0]
Statistical Analysis 4: Comparison: Placebo vs FP 100 µg BID; Test type: Superiority or Other; p = 0.459, ANCOVA; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-5.0 to 11.1]

8. Secondary Outcome: Number of Withdrawals Due to Lack of Efficacy Throughout the 12-week Treatment Period
Description: The number of participants whose primary reason for withdrawal from the study was due to lack of efficacy is presented together with p-values for the treatment comparisons.
Time Frame: Up to Week 12
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | FF 25 µg OD | FF 50 µg OD | FF 100 µg OD | FP 100 µg BID
Number analyzed (Participants) | 119 | 118 | 120 | 118 | 118
Participants | 42 | 16 | 23 | 21 | 19
Statistical Analysis 1: Comparison: Placebo vs FF 25 µg OD; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs FF 50 µg OD; Test type: Superiority or Other; p = 0.006, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p = 0.003, Fisher Exact
Statistical Analysis 4: Comparison: Placebo vs FP 100 µg BID; Test type: Superiority or Other; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the follow-up visit (up to 13 weeks).
Description: On-treatment SAEs and non-serious AEs are reported for members of the ITT Population, comprised of all participants who were randomized to treatment and received at least one dose of study medication.
Arm/Group | Placebo | FF 25 µg OD | FF 50 µg OD | FF 100 µg OD | FP 100 µg BID
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/118 | 1/120 | 1/118 | 0/118
Other Adverse Events (participants affected / at risk) | 20/119 | 27/118 | 20/120 | 29/118 | 24/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=119) | FF 25 µg OD (N=118) | FF 50 µg OD (N=120) | FF 100 µg OD (N=118) | FP 100 µg BID (N=118)
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=119) | FF 25 µg OD (N=118) | FF 50 µg OD (N=120) | FF 100 µg OD (N=118) | FP 100 µg BID (N=118)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 7 (9) | 1 (1) | 10 (12) | 5 (5)
Nasopharyngitis (Infections and infestations) | 4 (5) | 9 (12) | 4 (5) | 3 (3) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (9) | 1 (1) | 6 (8) | 5 (5)
Pharyngitis (Infections and infestations) | 4 (5) | 2 (2) | 7 (8) | 5 (5) | 1 (2)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 7 (10) | 4 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (8) | 2 (2) | 2 (2) | 4 (4)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.